CLINICAL TRIAL: NCT04533438
Title: The RhinAer Procedure for Treatment of CHronic RhInitis - A Prospective, MulticeNter Randomized ConTrolled TRial Comparing RhinAer to Sham Control (RHINTRAC)
Brief Title: RhinAer Procedure for Treatment of Chronic Rhinitis Study
Acronym: RHINTRAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aerin Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CTP1004
Record Dates: First submitted 2020-08-21; First posted 2020-08-31 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Chronic Rhinitis

STUDY DESIGN:
Intervention Model Description: 2:1 site-stratified randomization will be used to allocate participants to either the RhinAer procedure or treatment with the sham (control) procedure. Crossover within 30 days after 3- or 6-month follow-up visit.
Who Masked: Participant
Masking Description: Participant will be blinded to the study arm they are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- RhinAer Treatment (Active Comparator): The RhinAer procedure will be performed in the study clinic using the RhinAer Stylus and Aerin Console. The RhinAer Stylus is a disposable handheld device capable of delivering bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device. Participants will have the portion of the nasal cavity mucosa overlying the region of the posterior nasal nerve (the posterior middle meatus and posterior inferior turbinate) in both nostrils treated during a single study procedure session. Each nostril will be treated at 1, 2, 3, 4 or 5 nonoverlapping positions depending on the size of the target treatment area. Treatment settings to be used are temperature 60 °C, power 4 watts, treatment time 12 seconds, and cooling time 0 seconds
  Interventions: Device: RhinAer Stylus
- Control Treatment (Sham Comparator): The control treatment will be performed in the study clinic using the RhinAer Stylus while audible sounds that accurately simulate the Aerin Console's active treatment are produced even though RF energy is not being generated or delivered. All other aspects of the procedure will be the same as used for the active treatment, including administration of anesthetic agent(s).
  Interventions: Device: Sham

INTERVENTIONS:
Device: RhinAer Stylus — The RhinAer procedure will be performed in the study clinic using the RhinAer Stylus and Aerin Console. The RhinAer Stylus is a disposable handheld device capable of delivering bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device. Participants will have the portion of the nasal cavity mucosa overlying the region of the posterior nasal nerve (the posterior middle meatus and posterior inferior turbinate) in both nostrils treated during a single study procedure session.
  Arms: RhinAer Treatment
Device: Sham — The control treatment will be performed in the study clinic using the RhinAer Stylus while audible sounds that accurately simulate the Aerin Console's active treatment are produced even though RF energy is not being generated or delivered. All other aspects of the procedure will be the same as used for the active treatment, including administration of anesthetic agent(s).
  Arms: Control Treatment

SUMMARY:
The purpose of this study is to compare the RhinAer procedure with radiofrequency (RF) energy to sham procedure for treatment of chronic rhinitis.

DETAILED DESCRIPTION:
The purpose of this study is to compare the RhinAer procedure to treat tissue in the posterior nasal nerve area to improve symptoms in adults diagnosed with chronic rhinitis with a sham procedure that duplicates the actual procedure as closely as possible absent the delivery of radiofrequency (RF) energy to the nasal tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 85 years (inclusively).
2. Willing and able to provide informed consent.
3. Willing and able to comply with the subject-specific requirements outlined in the Study Protocol.
4. Seeking treatment for chronic rhinitis symptoms of at least 6 months duration and willing to undergo an office-based procedure.
5. Moderate to severe symptoms of rhinorrhea (rTNSS rating of 2 or 3 for rhinorrhea).
6. Mild to severe symptoms of nasal congestion (rTNSS rating of 1, 2 or 3 for congestion).
7. rTNSS ≥ 6.

Exclusion Criteria:

1. Anatomic obstructions that in the investigator's opinion limit access to the posterior nasal passage.
2. Altered anatomy of the posterior nose as a result of prior sinus or nasal surgery or injury.
3. Active nasal or sinus infection.
4. History of significant dry eye.
5. History of any of the following: chronic epistaxis, documented episodes of significant nose bleeds in the past 3 months, rhinitis medicamentosa, head or neck irradiation.
6. Have rhinitis symptoms only on a seasonal basis due to allergies.
7. Known or suspected allergies or contraindications to the anesthetic agents and/or antibiotic medications to be used during the study procedure session.
8. Known or suspected to be pregnant or is lactating.
9. Participating in another clinical research study.
10. Has any condition that predisposes to excessive bleeding.
11. Is taking anticoagulants (eg, warfarin, Plavix) or 325 mg aspirin that cannot be discontinued before the procedure.
12. Has previous procedure or surgery for chronic rhinitis.
13. Other medical conditions which in the opinion of the investigator would predispose the subject to poor wound healing, increased surgical risk, or poor compliance with the requirements of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Stolovitzky, MD, Principal Investigator — ENT of Georgia North; Mas Takashima, MD, Principal Investigator — The Sinus Center at Houston Methodist Hospital
Locations (13):
- United States (13):
  - Sacramento ENT (DaVinci Research), Roseville, California
  - Breathe Clear Institute, Torrance, California
  - ENT and Allergy Associates of Florida, Plantation, Florida
  - University of South Florida, Tampa, Florida
  - Piedmont ENT, Atlanta, Georgia
  - Rush University, Chicago, Illinois
  - Madison ENT, New York, New York
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Vanderbilt Asthma, Sinus & Allergy Program, Nashville, Tennessee
  - Texas Healthcare, Fort Worth, Texas
  - Fredericksburg ENT, Fredericksburg, Texas
  - ENT Associates of Texas (ENTtex), McKinney, Texas
  - Ogden Clinic, Ogden, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stolovitzky JP, Ow RA, Silvers SL, Bikhazi NB, Johnson CD, Takashima M. Effect of Radiofrequency Neurolysis on the Symptoms of Chronic Rhinitis: A Randomized Controlled Trial. OTO Open. 2021 Sep 10;5(3):2473974X211041124. doi: 10.1177/2473974X211041124. eCollection 2021 Jul-Sep. PMID 34527852
- [Result] Takashima M, Stolovitzky JP, Ow RA, Silvers SL, Bikhazi NB, Johnson CD. Temperature-controlled radiofrequency neurolysis for treatment of chronic rhinitis: 12-month outcomes after treatment in a randomized controlled trial. Int Forum Allergy Rhinol. 2023 Feb;13(2):107-115. doi: 10.1002/alr.23047. Epub 2022 Jul 5. PMID 35714267
- [Result] Takashima M, Stolovitzky JP, Ow RA, Silvers SL, McDuffie CM, Dean M, Sedaghat AR, Tajudeen BA. Temperature-controlled radiofrequency ablation for the treatment of chronic rhinitis: Two-year outcomes from a prospective multicenter trial. Int Forum Allergy Rhinol. 2024 Jul;14(7):1182-1194. doi: 10.1002/alr.23315. Epub 2024 Jan 24. PMID 38266636
- [Result] Stolovitzky JP, Ow RA, Silvers SL, Tajudeen BA, McDuffie CM, Dean M, Sedaghat AR, Phillips K, Takashima M. 3-Year Outcomes of Temperature-Controlled Radiofrequency Ablation of the Posterior Nasal Nerve in Patients With Chronic Rhinitis. Int Forum Allergy Rhinol. 2025 Sep;15(9):915-925. doi: 10.1002/alr.23577. Epub 2025 Apr 4. PMID 40183781

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at X academic medical centers and clinics between July 30, 2020 and December 29, 2020. The first participant was enrolled on July 31, 2020 and the last participant was enrolled in December 28,2020
Pre-assignment Details: There was no wash out or run in for this study
Period: Initial Enrollment
Arm/Group | RhinAer Treatment | Control Treatment
Started | 77 | 39
Completed | 77 | 39
Not Completed | 0 | 0
Period: Crossover Period
Arm/Group | RhinAer Treatment | Control Treatment
Started (The Crossover Period does not apply to subjects that were randomized to Rhinaer Treatment Arm) | 0 | 39
Completed | 0 | 28 (Subjects who received SHAM randomization were permitted to crossover to treatment are after 3M evaluation, only if they continued to meet the inclusion/exclusion criteria for the study. Subjects that did not meet inclusion/exclusion to crossover were exited as completed)
Not Completed | 0 | 11
Not completed — Did not meet Eligibility to Crossover | 0 | 11

BASELINE CHARACTERISTICS:
Groups:
- Active Treatment: Subjects randomized to receive the Rhinaer procedure
- Sham Control: Subjects randomized to receive the Sham Procedure
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Sham Control | Total
Number analyzed (Participants) | 77 | 39 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (14.8) | 57.8 (14.4) | 57.5 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 26 | 75
  Male | 28 | 13 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 69 | 36 | 105
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 0 | 2
Nasal Exam Turbinate Enlargement [Count of Participants; unit: Participants] | 16 | 8 | 24
Nasal Exam Nasal Polyps [Count of Participants; unit: Participants] | 3 | 0 | 3
Prior Nasal Surgery [Count of Participants; unit: Participants] | 27 | 13 | 40
rTNSS [Mean (Standard Deviation); unit: rTNSS Score] — TNSS is an instrument used to collect patient self-rated severity of nasal symptoms. The FDA cites this as a preferred measure of efficacy in trials of drug treatments for rhinitis. The total score is the sum of the 4 nasal symptom scores with a maximum TNSS of 12 indicating the most severe symptoms.
  Treatment Responder based on rTNSS improvement Individual participant success (responder) is defined as at least 30% improvement (decrease) in the rTNSS from baseline.
  rTNSS Score | 8.3 (1.9) | 8.2 (1.8) | 8.25 (1.85)
Medication Use - Antihistamines [Count of Participants; unit: Participants] | 56 | 28 | 84
Medication Use - Decongestants [Count of Participants; unit: Participants] | 22 | 10 | 32
Medication Use - Oral leukotriene inhibitors [Count of Participants; unit: Participants] | 4 | 3 | 7
Medication use - Intranasal steroid sprays [Count of Participants; unit: Participants] | 34 | 26 | 60
Medication Use -Intranasal anticholinergic sprays [Count of Participants; unit: Participants] | 19 | 8 | 27

OUTCOME MEASURES:

1. Primary Outcome: Reflective Total Nasal Symptom Score (rTNSS) Responder Rate
Description: TNSS is an instrument used to collect patient self-rated severity of nasal symptoms. 4 Symptoms (rhinorrhea, nasal congestion, nasal itching and sneezing) are reported with score of 0/absent; 1/mild; 2/moderate; 3/severe. The total score is the sum of the 4 nasal symptom scores with a maximum TNSS of 12 indicating the most severe symptoms. Treatment Responder based on rTNSS improvement Individual participant success (responder) is defined as at least 30% improvement (decrease) in the rTNSS from baseline.
  For this protocol patients had to meet inclusion criteria of rTNSS rating of 2 or 3 for Rhinorrhea; rTNSS rating of 1, 2 or 3 for Congestion; and total rTNSS score >/= 6 at baseline
Time Frame: 3 months visit following the study procedure.
Measure: Count of Participants; unit: Participants
Groups:
- Active Treatment: Subject randomized who received Rhinaer Treatment
- Sham Control: Subject randomized who received Sham Treatment
Arm/Group | Active Treatment | Sham Control
Number analyzed (Participants) | 77 | 39
Participants | 52 | 16

2. Secondary Outcome: Reflective Total Nasal Symptom Score (rTNSS) Mean Change
Description: The Reflective Total Nasal Symptom Score (rTNSS) is a patient self reported questionnaire of four nasal symptoms: rhinitis, nasal congestion, nasal itching and sneezing. Patients will report their symptoms reflected or felt over the last 12 hours. Total scores can range from 0 to 12. A higher score indicates increased symptom severity.
  This study will measure the mean change in rTNSS from baseline to 3 months after the procedure.
Time Frame: Change from Baseline to 3 months following the study procedure.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Treatment | Sham Control
Number analyzed (Participants) | 77 | 39
score on a scale | -3.6 [-4.2 to -3.0] | -2.2 [-3.2 to -1.3]

3. Secondary Outcome: Reflective Total Nasal Symptom Score (rTNSS) Mean Change
Description: The Reflective Total Nasal Symptom Score (rTNSS) is a patient self reported questionnaire of four nasal symptoms: rhinitis, nasal congestion, nasal itching and sneezing. Patients will report their symptoms reflected or felt over the last 12 hours. Total scores can range from 0 to 12. A higher score indicates increased symptom severity.
Time Frame: Change from Baseline to 12 months following the study procedure.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Combined Active and Sham Treatment Group: Patient disposition, active treatment group and including crossover of the index sham-control arm to active treatment at 3 months
Arm/Group | Combined Active and Sham Treatment Group
Number analyzed (Participants) | 88
score on a scale | -4.8 [-5.5 to -4.1]

4. Secondary Outcome: Percentage of Participants With Treatment Related Events (Safety)
Description: Characterizing the type and frequency of adverse events reported. Subjects will be asked about possible side effects or adverse experiences related to the study procedure at each follow up visit. All events will be documented and identified as to its relationship and level of relatedness to the study device and/or study procedure. Date of onset, severity, duration and outcome will be documented.
Time Frame: At or following the study procedure up to to 3 months.
Measure: Count of Participants; unit: Participants
Groups:
- Active Treatment: Subject randomized who received Rhinaer Procedure
- Sham Control: Subject randomized who received Sham Procedure
Arm/Group | Active Treatment | Sham Control
Number analyzed (Participants) | 77 | 39
Participants
  Severe Nasal Soreness/Pain | 1 | 0
  Increased Nasal Congestion at 1 month | 1 | 0
  Mild nasal bleeding immediate post procedure | 0 | 1

5. Other Pre Specified Outcome: Nasal Status Assessment
Description: The Nasal Status Assessment is an evaluation, performed by a physician, of 10 specified physical or intranasal findings. Each finding is ranked in severity from Not Present to Severe. Each component of the assessment will be summarized.
Time Frame: Baseline, 1 month, 3 months and 6 months following the study procedure
Measure: Number; unit: participants
Arm/Group | Active Treatment | Sham Control
Number analyzed (Participants) | 77 | 39
participants
  Significant Dry Eye | 1 | 0
  Soreness, Pain | 3 | 4

ADVERSE EVENTS:
Time Frame: 3 months
Description: AE- any untoward medical occurrence in a subject SAE-an AE that: led to death, led to serious deterioration in the health, resulted in a life-threatening illness or injury, resulted in permanent impairment of body structure or body function, required hospitalization or prolongation of existing hospitalization, resulted in medical or surgical intervention to prevent permanent impairment, led to fetal distress, fetal death, a congenital abnormality, or birth defect
Groups:
- RhinAer Treatment: The RhinAer procedure will be performed in the study clinic using the RhinAer Stylus and Aerin Console. The RhinAer Stylus is a disposable handheld device capable of delivering bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device. Participants will have the portion of the nasal cavity mucosa overlying the region of the posterior nasal nerve (the posterior middle meatus and posterior inferior turbinate) in both nostrils treated during a single study procedure session. Each nostril will be treated at 1, 2, 3, 4 or 5 nonoverlapping positions depending on the size of the target treatment area. Treatment settings to be used are temperature 60 °C, power 4 watts, treatment time 12 seconds, and cooling time 0 seconds RhinAer Stylus: The RhinAer procedure will be performed in the study clinic using the RhinAer Stylus and Aerin Console. The RhinAer Stylus is a disposable handheld device capable of delivering bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device. Participants will have the portion of the nasal cavity mucosa overlying the region of the posterior nasal nerve (the posterior middle meatus and posterior inferior turbinate) in both nostrils treated during a single study procedure session.
Arm/Group | RhinAer Treatment | Control Treatment
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/39
Other Adverse Events (participants affected / at risk) | 7/77 | 1/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RhinAer Treatment (N=77) | Control Treatment (N=39)
Nasal Bleeding (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) — Nasal Bleeding
Nasal Congestion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) — Nasal Congestion
Headache (Nervous system disorders) | 1 (1) | 1 (1) — Headache
Vasovagal Reaction (Nervous system disorders) | 1 (1) | 0 (0) — Vasovagal Reaction

LIMITATIONS AND CAVEATS:
Patients with a predisposition to poor wound healing were excluded from this trial, and therefore, the results may not be applicable to this patient population. Investigators were not blinded. The rTNSS used in endpoint evaluation was reported by the blinded patient, mitigating the risk of bias. Pain VAS was completed by the blinded patients. Allergy testing not required and relative efficacy by rhinitis subtype could not be compared. Medication use was not controlled

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT04533438/Prot_SAP_000.pdf